CLINICAL TRIAL: NCT05155228
Title: Evaluation of the Attachment, Regulation and Competency (ARC) Framework for the Treatment of Complex Trauma in Children
Brief Title: The Attachment, Regulation and Competency (ARC) Framework
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Justice Resource Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JRI 2016-03
Record Dates: First submitted 2017-03-24; First posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: Posttraumatic Stress Disorder; Developmental Trauma Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Mental Competency; Therapeutics

STUDY DESIGN:
Intervention Model Description: The Attachment, Regulation and Competency (ARC) Framework is an attachment focused model designed specifically for trauma-impacted children that incorporates principles of the following theoretical orientations: 1) developmental theory; 2) family systems theory; and 3) strengths-based approaches. The central goals of the ARC framework are to (a) support caregiving systems and enhance caregiver-child relationships ("Attachment"), (b) support children in developing the skills and tolerance for connecting to, identifying, and sharing internal experience and managing emotional and physiological states ("Regulation"), (c) build key capacities associated with resilience including the ability to engage in problem-solving and a positive / effective sense of self ("Competency"), and (d) process traumatic experiences.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Attachment Regulation and Competency (Experimental): Weekly individual psychotherapy for 24 weeks using the Attachment Regulation and Competency intervention.
  Interventions: Behavioral: Attachment Regulation and Competency
- Treatment as usual (Active Comparator): Weekly individual psychotherapy for 24 weeks.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Attachment Regulation and Competency — Trauma informed psychotherapy intervention for children with a history of exposure to trauma and their caregivers.
  Arms: Attachment Regulation and Competency
Behavioral: Treatment as usual — Supportive psychotherapy
  Arms: Treatment as usual

SUMMARY:
This study evaluates the effectiveness of the Attachment Regulation and Competency (ARC) treatment framework in comparison to treatment as usual for reducing symptoms of PTSD and Developmental Trauma Disorder among children ages 8 to 16 with a history of exposure to multiple traumatic events.

DETAILED DESCRIPTION:
The primary goal of this project is to expand the knowledge base in the field of trauma informed interventions by addressing current gaps in the evidence base through: a) evaluation of the efficacy of an innovative intervention designed specifically for children who experience complex trauma and their caregivers, thereby evaluating strategies that are most effective, and b) examining how ARC promotes protective factors (self-regulation, caregiver wellness), thereby supporting the health and well-being of complexly traumatized children and their families. The overall purpose of the randomized controlled trial (RCT) is to examine the effectiveness of ARC on the range of developmental disruptions and clinical symptoms that represent complex trauma, as well as its utility for increasing the adaptive functioning of children and families. In particular it is necessary to determine: 1) if ARC will demonstrate effectiveness in reducing sequelae of complex trauma as determined by a scientifically rigorous randomized control trial study design; 2) the extent to which ARC positively impacts resiliency factors (self-regulation, executive functioning, caregiver wellness), thereby serving to moderate or mediate change in symptoms and functioning; and 3) the impact of ARC across multiple levels of the family ecology, including the child, the caregiver-child relationship (i.e., attachment) and caregiver stress and wellness.

The specific objectives of this research project are the following:

1. Recruit 182 children ages 8 to 16 with complex trauma and their adult caregivers, from clinical samples of children actively seeking treatment for mental health disorders and related difficulties from three community based outpatient clinics in the Commonwealth of Massachusetts.
2. Conduct comprehensive, clinical interviews with participants and their caregivers to assess sequelae of complex trauma, to determine underlying resiliency factors and to gather information regarding trauma exposure history, over four study time points (pre-, mid-, and post-treatment and 6-month follow up).
3. Deliver 24 sessions of once weekly ARC or TAU over a 6-month intervention period.
4. Evaluate the efficacy of ARC and TAU using a variety of sophisticated statistical methods, such as growth curve modeling, multivariate analyses, and hierarchical linear regression analyses.
5. Disseminate findings to: 1) the academic community via presentations at professional conferences and publications of data in peer reviewed journals; 2) the public, via the Trauma Center website, which received over 600,000 visitors in 2012, with 1,161,451 downloads of our manuscripts and resources for providers, consumers and state service agencies; and 3) the National Child Traumatic Stress Network (NCTSN) and Complex Trauma Treatment Network (CTTN) at annual network meetings, via their websites and through ongoing collaborations with partner network sites across the country.

ELIGIBILITY:
Inclusion Criteria.

1. DTD diagnosis as measured by the DTD interview (using standard scoring criteria) or partial PTSD diagnosis as measured by the CAPS.
2. A history of at least two forms of trauma, at least one of which must be interpersonal in nature (sexual, physical or psychological maltreatment, neglect, abandonment or impaired caregiving) as indicated on the Trauma History Profile (THP).

Exclusion Criteria.

1. Serious illness that is not stabilized.
2. GAF < 40.
3. Past diagnosis of autism spectrum disorder, mental retardation, or schizophrenia.
4. Current psychotic disorder or established organic impairment (e.g., TBI).
5. Active suicidal risk, self-mutilation or homicidal behavior toward others within the past 3 months, as judged by the PI.
6. Previous ARC treatment.
7. Any other condition that might interfere with the person's capacity to give informed consent, or to adhere to the study protocol.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Change in baseline symptoms of PTSD at up to 24 weeks of treatment and 6-month follow up per the Clinician Administered PTSD Scale for Children and Adolescents, DSM 5 (CAPS-CA-DSM5) | Change from baseline PTSD symptom severity at up to 24 weeks of treatment and 6-month follow up.
  The Clinician Administered PTSD Scale for Children and Adolescents, DSM 5 (CAPS-CA-DSM5) is a clinical research interview assessing the severity and frequency of DSM 5 symptoms of posttraumatic stress disorder over the previous month. The CAPS yields a total severity score based on assessment of 20 symptoms of PTSD that can range from 0 to 80, with higher scores indicating a greater severity of PTSD symptoms.
Change in baseline symptoms of Developmental Trauma Disorder (DTD) at up to 24 weeks of treatment and 6-month follow up | Change from baseline DTD symptom severity at up to 24 weeks of treatment and 6-month follow up.
  The Developmental Trauma Disorder Structured Interview (DTD-SI) is a clinician-administered semi-structured diagnostic interview designed for a parent or other primary caregiver of a child 8 to 17 years old to describe problems the child has in three categories of dysregulation: (1) Affective and Physiological, (2) Attentional and Behavioral, (3) Self and Relational. Questions and interviewer ratings parallel those of the K-SADS. The DTD-SI yields a total symptom score ranging from 0 to 25, with higher scores indicating greater severity of DTD symptoms.

SECONDARY OUTCOMES:
UCLA Posttraumatic Stress Disorder -Reaction Index for DSM 5 (PTSD-RI-5) | Change from baseline PTSD symptom severity at up to 12-weeks of treatment, up to 24 weeks of treatment and 6-month follow up.
  The UCLA Posttraumatic Stress Disorder -Reaction Index for DSM 5 (PTSD-RI-5) includes 31 items which map closely to the DSM 5 symptom criteria, yields a total score ranging from 0 to 124 with higher scores indicating more severe symptoms of PTSD, and provides clinical cut-off scores that can be used to measure severity of PTSD symptoms.
Child Behavior Checklist (CBCL) | Change from baseline in internalizing and externalizing problems at up to 12 weeks of treatment, up to 24 weeks of treatment, and 6-month follow up.
  The Child Behavior Checklist is a 113 item, caregiver report of aggressive behavior, internalizing and externalizing symptoms, and dysregulation for youth ages 6-18 years of age, yielding nine syndrome scales and six DSM-oriented scales. The CBCL yields a Total Score ranging from 0 to 226, with higher scores indicating more severe emotional and behavioral problems.
Behavior Rating Inventory of Executive Function - Parent Report (BRIEF-PR) | Change from baseline in executive dysfunction at up to 12 weeks of treatment, up to 24 weeks of treatment and 6-month follow up.
  The Behavior Rating Inventory of Executive Function - Parent Version (BRIEF-PR) assesses various domains of executive function, including two broad scales; behavioral regulation (composed of inhibition, shifting and emotional control) and metacognition (composed of initiation, working memory, planning/organization, monitoring and organization of materials) and a global EF composite score. This 86-item measure yields a Global Executive Function score ranging from 0 to 176, with higher scores indicating poorer executive functions.
Trauma Symptom Checklist for Children (TSCC) | Change from baseline in symptoms of dissociation at up to 12 weeks of treatment, up to 24 weeks of treatment, and 6-month follow up.
  The Trauma Symptom Checklist for Children (TSCC) is 54-item child report for children ages 8-16 years to assess distress and related symptoms of trauma, including subscales for PTSD symptoms, dissociation, depression, anxiety, and sexual concerns. Scores for each subscale range from 9 to 36, with higher scores indicating greater symptom severity in a given domain.
NIH Toolbox for the Assessment of Neurological and Behavioral Function, Cognition Domain | Change from baseline in executive function at up to 12 weeks of treatment, up to 24 weeks of treatment and 6-month follow up.
  state-of-the-art computer-administered measures of cognitive function for use with subjects aged 3-85 years:
  (a) Flanker Task: measure of inhibitory control in the context of selective visual attention. Youth indicate the left-right orientation of a stimulus (fish or arrow) while ignoring incongruent flankers (oriented the opposite way), (b) DCCS: measures cognitive flexibility. Youth sort stimuli using to a cued rule (shape/color), and (c) List Sorting: measures working memory, requiring maintenance/manipulation of information.

OTHER OUTCOMES:
Behavioral and Emotional Rating Scale, Second Edition (BERS-2) | Change from baseline in resilience at up to 12 weeks of treatment, up to 24 weeks of treatment and 6-month follow up.
  The Behavioral and Emotional Rating Scale, Second Edition (BERS-2) is parent report measure assessing resiliency by measuring youth competencies, including interpersonal and intrapersonal strength, family involvement, school functioning, affective strength and career strength. The BERS-2 yields a total score ranging from 0 to 171 with higher scores indicating greater resilience.
Emotion Regulation Checklist (ERC) | Change from baseline in emotion regulation at up to 12 weeks of treatment, up to 24 weeks of treatment and 6-month follow up.
  Emotion Regulation Checklist (ERC) is a parent-report measure of child emotion regulation, emotional lability and negative affect. The Emotion Regulation subscale is comprised of 8 items which measure empathy, self-awareness of emotion, and appropriateness of emotional displays. Scores on the Emotion Regulation subscale range from 8 to 32, with higher scores reflecting greater regulatory abilities. The Lability/Negativity subscale reflects temperament-related behavior such as mood swings, angry reactivity, and intensity of positive and negative emotions, with scores ranging from 16 to 64, with higher scores indicating greater emotional negativity and lability.
Brief Symptom Inventory (BSI) | Change from baseline in caregiver mental health symptoms at up to 12 weeks of treatment, up to 24 weeks of treatment and 6-month follow up.
  The Brief Symptom Inventory (BSI) is a 53 item measure assessing nine symptom dimensions including Somatization, Obsession-Compulsion, Interpersonal Sensitivity, Depression, Anxiety, Hostility, Phobic anxiety, Paranoid ideation and Psychoticism in adults and will be used to assess caregiver mental health symptoms. Scores range from 0 to 216 with greater scores indicating greater mental health problems.

CONTACTS AND LOCATIONS:
Overall Officials: Hilary B Hodgdon, Ph.D., Principal Investigator — Trauma Center at JRI
Locations (1):
- Trauma Center at JRI, Brookline, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
At this time IPD will not be shared with other researchers.